CLINICAL TRIAL: NCT01694875
Title: Clinical Evaluation of the APTIMA® HPV 16 18/45 Genotype Assay on the PANTHER® System in Women With ASC-US Pap Test Results and in Women 30 Years of Age or Older With Negative Pap Test Results Using ThinPrep Pap Test Specimens
Brief Title: Clinical Evaluation of the APTIMA® HPV 16 18/45 Genotype Assay on the PANTHER® System
Status: Completed | Type: Observational
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: HPVGPS-US12-001
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Human Papillomavirus Infection
Keywords: cervix cancer; HPV; APTIMA
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment
  Interventions: Device: APTIMA HPV Assay

INTERVENTIONS:
Device: APTIMA HPV Assay — In Vitro Diagnostics Assay

SUMMARY:
The objective of the clinical study is to evaluate the AHPV-GT Assay using the PANTHER System in cervical cancer screening.

This objective will be accomplished in the ASC-US Study by evaluating the performance characteristics of the AHPV-GT Assay using the PANTHER System in a sample population of women with ASC-US Pap test results who were 21 years of age or older ("≥21 years of age") at the time of their Pap visit. For the Adjunct Study, this objective will be accomplished by evaluating the ability of the AHPV-GT Assay using the PANTHER System to identify women at increased risk of cervical disease in a sample population of women with negative (NILM)cytology results who were ≥30 years of age at the time of their Pap visit.

ELIGIBILITY:
Inclusion Criteria:

Subjects who were previously enrolled into the prospective, multicenter US clinical study for the APTIMA HPV Assay on the TIGRIS System (protocol 2007HPVASCUS30) will be eligible for inclusion in the study of the AHPV-GT Assay using the PANTHER System described in this protocol. All evaluable ASC-US Study subjects ≥21 years of age will be eligible for inclusion.

Evaluable Adjunct Study subjects ≥30 years of age will be eligible if the following criteria are met:

* the subject attended the colposcopy visit, or
* the subject did not attend the colposcopy visit but the referral Pap sample had a positive APTIMA HPV Assay result in the APTIMA HPV Assay TIGRIS System study (protocol 2007HPVASCUS30) or in the APTIMA HPV Assay PANTHER System study (protocol AHPVPS-US11-003).

Exclusion Criteria:

Eligible subjects will be excluded if they do not have an evaluable sample. This may be due to insufficient volume or because the sample was deemed unsuitable for testing (eg, stored under unacceptable conditions).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples from subjects who attended colposcopy from the Adjunct Study and subjects who had positive APTIMA HPV Assay results in the APTIMA HPV Assay TIGRIS System Study or the APTIMA HPV Assay PANTHER System Study.
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reid, PhD, Study Director — Gen-Probe, Incorporated
Locations (3):
- United States (3):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Laboratory Corporation of America, Burlington, North Carolina
  - Molecular Pathology Laboratory Network, Inc, Maryville, Tennessee